CLINICAL TRIAL: NCT03032406
Title: CLEVER Pilot Trial: A Phase II Pilot Trial of HydroxyChLoroquine, EVErolimus or the Combination for Prevention of Recurrent Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 24116
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Results first posted 2025-03-05 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer Stage IIB
MeSH Terms: conditions — Breast Neoplasms | interventions — Hydroxychloroquine; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- HCQ alone (Arm A) (Experimental)
  Interventions: Drug: Hydroxychloroquine
- EVE alone (Arm B) (Experimental)
  Interventions: Drug: Everolimus
- combination HCQ and EVE (Arm C+D) (Experimental)
  Interventions: Drug: Hydroxychloroquine; Drug: Everolimus

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine
  Arms: HCQ alone (Arm A); combination HCQ and EVE (Arm C+D)
Drug: Everolimus — Everolimus
  Arms: EVE alone (Arm B); combination HCQ and EVE (Arm C+D)

SUMMARY:
To evaluate the feasibility of administering HCQ, EVE or the combination in patients who have completed primary therapy for breast cancer and harbor bone marrow disseminated tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed, primary, invasive breast cancer diagnosed within 5 years of study entry.
* Qualifying risk status, at diagnosis utilizing receptor testing by

ASCO/CAP guidelines, meeting one of the following:

* Histologically positive axillary lymph nodes
* Primary tumor that is ER/PR/Her2 negative
* Primary tumor that is ER+/Her2 negative/Lymph node negative with Breast Cancer Recurrence Score of ≥ 25 per the Genomic Health Oncotype DX breast cancer test
* Evidence of residual disease in the breast on pathological assessment after neoadjuvant chemotherapy.
* Patients must have completed all primary therapy (definitive surgery, (neo)adjuvant chemotherapy adjuvant radiation and/or Her2-directed therapy) for the index malignancy at least 4 weeks prior to study entry. All prior treatment-related toxicity must be resolved prior to study enrollment. Concurrent receipt of adjuvant endocrine and bone modifying agents is allowed per standard of care guidelines.
* Bone marrow aspirate after completion of therapy demonstrates detectable DTCs (via IHC)
* No evidence of recurrent local or distant breast cancer by physical examination, blood tests (CBC, LFTs, Alk Phos), or symptom-directed imaging, per NCCN guidelines.
* Age ≥ 18 years
* ECOG performance status 2
* No contraindications to the study medications or uncontrolled medical illness.
* Adequate bone marrow function as shown by: ANC ≥ 1.5 x 109/L, Platelets ≥ 100 x 109/L, Hb >9 g/dL
* Adequate liver function as shown by: Serum bilirubin ≤ 1.5 x ULN, ALT and AST ≤ 2.5 x ULN, and INR ≤1.5
* Anticoagulation is allowed if target INR ≤ 1.5 on a stable dose of warfarin or on a stable dose of anticoagulant for >2 weeks at time of randomization. For patients on therapeutic anti-coagulants, medication must be clinically held peri-procedure (bone marrow aspirate) per standard clinical management.
* Adequate renal function: serum creatinine ≤ 2.0 x ULN or creatinine clearance (CrCl) ≥ 30mL/min obtained within 28 days prior to registration. A calculated creatinine clearance by Cockcroft-Gault Formula is acceptable in lieu of a measured value.
* Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
* Ability to provide informed consent

Exclusion criteria

* Concurrent enrollment on another investigational therapy
* Prior treatment with an mTOR inhibitor (sirolimus, temsirolimus, everolimus).
* Known hypersensitivity to Everolimus or other rapamycins (sirolimus, temsirolimus) or to its excipients.
* Patients receiving chronic, high dose systemic treatment with corticosteroids defined as: chronic use of cortisone >50mg; hydrocortisone >40mg, prednisone >10mg, methylprednisone >8mg or dexamethasone > 1.5mg; or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study including: Symptomatic congestive heart failure of New York heart Association Class III or IV Unstable angina pectoris, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease Severely impaired lung function with a previously documented spirometry and DLCO that is 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air Uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN Active (acute or chronic) or uncontrolled severe infections Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis A known history of HIV seropositivity as reported by the patient Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of EVE (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection) Patients with an active, bleeding diathesis Active or latent, untreated Hepatitis B or C. A detailed assessment of Hepatitis B/C medical history and risk factors must be done at screening for all patients. HBV DNA and HCV RNA PCR testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV/HCV infection.
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. If barrier contraceptives are being used, these must be continued throughout the trial and for 8 weeks after stopping study drug, by both sexes. Hormonal contraceptives are not acceptable as a sole method of contraception. (Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to administration of EVE.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2026-01-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Angela DeMichele, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] DeMichele A, Clark AS, Shea E, Bayne LJ, Sterner CJ, Rohn K, Dwyer S, Pan TC, Nivar I, Chen Y, Wileyto P, Berry LR, Deluca S, Savage J, Makhlin I, Pant DK, Martin H, Egunsola A, Mears N, Goodspeed BL, Chislock EM, Graves J, Wang J, Shih N, Belka GK, Berry D, Nayak A, Feldman M, Chodosh LA. Targeting dormant tumor cells to prevent recurrent breast cancer: a randomized phase 2 trial. Nat Med. 2025 Oct;31(10):3464-3474. doi: 10.1038/s41591-025-03877-3. Epub 2025 Sep 2. PMID 40897974

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The target accrual was originally 60; but due to slow enrollment caused by the Covid-19 pandemic, the target enrollment was modified and study enrollment was completed after each 15 patients became evaluable in each treatment group (Arm A, Arm B, and Arm C+D combined). We hit this target after a total of 51 patients were enrolled and treated. 53 patients were randomized but two dropped out before receiving an intervention.
Groups:
- Combination HCQ and EVE (Arm C); Combination HCQ and EVE 3-mo Delay (Arm D): Hydroxychloroquine: Hydroxychloroquine
  Everolimus: Everolimus
Period: Overall Study
Arm/Group | HCQ Alone (Arm A) | EVE Alone (Arm B) | Combination HCQ and EVE (Arm C) | Combination HCQ and EVE 3-mo Delay (Arm D)
Started | 15 | 15 | 8 | 15
Completed | 15 | 15 | 8 | 13
Not Completed | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The rationale for combining Arms C+D for certain analyses is because these arms are the same intervention- Arm D was just delayed. These arms are consistent with the protocol and randomization engine.
Groups:
- Total: Total of all reporting groups
Arm/Group | HCQ Alone (Arm A) | EVE Alone (Arm B) | Combination HCQ and EVE (Arm C+D) | Total
Number analyzed (Participants) | 15 | 15 | 23 | 53
Age, Continuous [Median (Full Range); unit: years] | 50.0 [31 to 66] | 45 [33 to 64] | 55 [34 to 73] | 50 [31 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 23 | 53
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 14 | 22 | 51
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 4 | 6
  White | 15 | 13 | 19 | 47
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Menopausal Status [Count of Participants; unit: Participants]
  Premenopausal | 4 | 8 | 5 | 17
  Postmenopausal | 11 | 7 | 18 | 36
Treatment [Count of Participants; unit: Participants]
  Adjuvant Chemotherapy | 6 | 6 | 13 | 25
  Neoadjuvant Chemotherapy | 8 | 9 | 9 | 26
  No Chemotherapy | 1 | 0 | 1 | 2
Receptor Subtype [Count of Participants; unit: Participants]
  ER+/Her2- | 6 | 3 | 7 | 16
  ER+/Her2+ | 1 | 2 | 1 | 4
  TNBC | 8 | 10 | 13 | 31
  ER-/Her2+ | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Feasibility: Number of Participants Who Completed 6 Cycles of Protocol Treatment Without Grade 3 or 4 Toxicity
Description: For the primary endpoint of feasibility, we employed ongoing Bayesian toxicity monitoring after every 3 participants completed cycle 6, assuming a Beta (1,2) prior, equivalent to one DLT observed in 3 treated participants. Early termination of a treatment arm for toxicity (non-feasibility) would occur if the posterior probability that the toxicity rate exceeds the target maximum of 30% was greater than 75%. Trial enrollment and conduct was significantly impacted by the COVID pandemic, including shortage of HCQ and inability of enrolled patients to travel. To address this, we amended the protocol to allow study Arms C and D to be combined for feasibility assessment, given that the investigational treatment was the same in the two arms, enabling enrollment to be halted when the sample size needed for feasibility assessment was complete for all study treatments. Toxicity was assessed using CTCAE v4.0.
Time Frame: 3 years
Population: Fifty-one of 53 participants were evaluable for the primary endpoint (excluding the 2 patients randomized to Arm D who withdrew during observation).
Measure: Count of Participants; unit: Participants
Arm/Group | HCQ Alone (Arm A) | EVE Alone (Arm B) | Combination HCQ and EVE (Arm C+D)
Number analyzed (Participants) | 15 | 15 | 21
Participants
  Feasible | 15 | 15 | 20
  Non-Feasible | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Patients were assessed for adverse events (AE) on Day 1 of each cycle. Follow-up continued every 6 months for 3 years from the completion of study therapy, including remote follow-up during COVID and for patients at a geographical distance from the study center. On Day 1 and D15 of first two cycles, then Day 1 of remaining cycles, and up to 30 days from completion of treatment.
Description: The rationale for combining Arms C+D for certain analyses is because these arms are the same intervention- Arm D was just delayed. These arms are consistent with the protocol and randomization engine.
Arm/Group | HCQ Alone (Arm A) | EVE Alone (Arm B) | Combination HCQ and EVE (Arm C+D)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/21
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/15 | 2/21
Other Adverse Events (participants affected / at risk) | 15/15 | 15/15 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HCQ Alone (Arm A) (N=15) | EVE Alone (Arm B) (N=15) | Combination HCQ and EVE (Arm C+D) (N=21)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cellulitis of arm (Infections and infestations) | 0 | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HCQ Alone (Arm A) (N=15) | EVE Alone (Arm B) (N=15) | Combination HCQ and EVE (Arm C+D) (N=21)
Diarrhea (Gastrointestinal disorders) | 12 | 5 | 14
Discomfort (Gastrointestinal disorders) | 9 | 8 | 13
Nausea (Gastrointestinal disorders) | 10 | 7 | 9
Liver function abnormalities (transaminitis) (Gastrointestinal disorders) | 7 | 3 | 15
Mucositis/oral pain (Gastrointestinal disorders) | 0 | 11 | 14
Anorexia/Weight loss (Gastrointestinal disorders) | 3 | 5 | 8
Constipation (Gastrointestinal disorders) | 4 | 6 | 4
Neutrophil count decreased (Blood and lymphatic system disorders) | 5 | 6 | 6
Leukocyte count decreased (Blood and lymphatic system disorders) | 4 | 6 | 7
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 6
Platelet count decreased (Blood and lymphatic system disorders) | 1 | 7 | 3
Visual changes (Nervous system disorders) | 5 | 2 | 10
Headache (Nervous system disorders) | 3 | 6 | 6
Dizziness (Nervous system disorders) | 4 | 0 | 3
Muscle weakness, limb (Nervous system disorders) | 2 | 0 | 5
CPK increased (Nervous system disorders) | 2 | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 5
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Electrolyte abnormalities (Renal and urinary disorders) | 0 | 7 | 11 — Laboratory Abnormalities
Hyperglycemia (Endocrine disorders) | 2 | 3 | 3 — Laboratory Abnormalities
Elevated lipids (Cardiac disorders) | 2 | 10 | 13 — Laboratory Abnormalities
Elevated creatinine (Renal and urinary disorders) | 4 | 0 | 5 — Laboratory Abnormalities
Fatigue (General disorders) | 6 | 7 | 11
SkinRash/Discomfort (Skin and subcutaneous tissue disorders) | 3 | 8 | 12
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 4

LIMITATIONS AND CAVEATS:
The results are limited by the small study sample size, low event rates, and lack of a placebo control.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/06/NCT03032406/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT03032406/SAP_003.pdf
  • Informed Consent Form (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT03032406/ICF_002.pdf